CLINICAL TRIAL: NCT02516202
Title: The Vaginal Health Trial - Effects of Vaginal Estradiol Tablet and Moisturizing Gel on Postmenopausal Vaginal Symptoms
Brief Title: The Vaginal Health Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: University of Minnesota (Other); Massachusetts General Hospital (Other); University of California, San Diego (Other); University of Washington (Other); Kaiser Permanente (Other)
Responsible Party: Principal Investigator, Katherine Guthrie, Principal Investigator, Fred Hutchinson Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MsFLASH 05; 8378 (Other: FHCRC IRB)
Record Dates: First submitted 2015-08-03; First posted 2015-08-05 (Estimated); Results first posted 2018-07-12 (Actual); Last update posted 2018-07-12 (Actual); Status verified 2018-06

CONDITIONS: Atrophy of Vagina; Menopause; Dyspareunia (Female)
MeSH Terms: conditions — Dyspareunia | interventions — Estradiol; segesterone acetate and ethinyl estradiol vaginal system

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (3):
- Vagifem (Active Comparator): One hundred participants will be randomized into the Vagifem® 'active' arm. These women will receive a bottle of Vagifem® tablets (estradiol 10 mcg). One tablet is to be inserted vaginally daily for 2 weeks, then 2 days/week for the remaining 10 weeks of the study.
  Vagifem® tablets contain 10.3 mcg of estradiol hemihydrate equivalent to 10 mcg of estradiol. The excipient (inactive) ingredients are hypromellose, lactose monohydrate, maize starch, and magnesium stearate. Vagifem® comes as a small white film-coated tablet. The coating is made of hypromellose and polyethylene glycol.
  A placebo gel visually similar to Replens composed of inert hydroxyethylcellulose gel (pH adjusted) applied every 3 days over entire 12 weeks.
  Interventions: Drug: Vagifem; Other: Placebo gel
- Replens (Active Comparator): One hundred participants will be randomized into the Replens® 'active' arm. These women will receive a tube containing Replens® vaginal gel, with 2.5 gm applied vaginally every 3 days over 12 weeks.
  Replens® is a bioadhesive polycarbophil-based moisturizing vaginal gel containing; purified water (vehicle humectant), glycerin (moisturizer), mineral oil (as a moisturizer), polycarbophil and carbomer homopolymer type B (allow the product to stick to the vaginal wall), hydrogenated palm oil glyceride (moisturizer), sorbic acid (preservative, antimicrobial), methylparaben, sodium hydroxide (adjusts pH of product so it is suitable for vaginal use).
  A placebo tablet visually identical to Vagifem® is inserted daily for 2 weeks, then 2 days/week for remaining 10 weeks.
  Interventions: Device: Replens; Other: Placebo tablet
- Placebo (Placebo Comparator): One hundred participants will be randomized into the 'placebo' arm of the study. This arm is comprised of two placebo preparations; placebo tablet and placebo gel applied on the same schedule as 'active' arms.
  The placebo tablet coating and excipient ingredients will be the same as are used for Vagifem®; the coating is made of hypromellose and polyethylene glycol and the excipient (inactive) ingredients are hypromellose, lactose monohydrate, maize starch, and magnesium stearate.
  Placebo gel. The product is an inert hydroxyethylcellulose gel (pH adjusted).
  Interventions: Other: Placebo tablet; Other: Placebo gel

INTERVENTIONS:
Drug: Vagifem — One tablet is to be inserted vaginally daily for 2 weeks, then 2 days/week for the remaining 10 weeks of the study.
  Other Names: vaginal estradiol
  Arms: Vagifem
Device: Replens — 2.5 gm to be applied vaginally every 3 days over 12 weeks.
  Other Names: non-hormonal hydrophilic non-prescriptive vaginal gel
  Arms: Replens
Other: Placebo tablet — Dispensed in visually identical bottle and tablet form to Vagifem.
  Arms: Placebo; Replens
Other: Placebo gel — Dispensed in visually identical tube and gel form to Replens.
  Arms: Placebo; Vagifem

SUMMARY:
This is a new application from the Menopause Strategies: Finding Lasting Answers for Symptoms and Health (MsFLASH) Clinical Trials network. Here we propose to conduct a large multicenter trial comparing two common treatments, a vaginal hormone tablet and an over-the-counter gel, with placebo to evaluate their effects on bothersome vaginal symptoms and sexual function, and to create a biorepository of specimens for future translational, mechanistic research on the etiology of vaginal symptoms.

DETAILED DESCRIPTION:
The Menopause Strategies: Finding Lasting Answers for Symptoms and Health (MsFLASH) Clinical Trials network was established in 2009. By the end of 2014, the network completed 4 clinical trials testing 7 interventions in approximately 1000 women ages 40-62 with vasomotor (VMS) and other menopause symptoms.

The current trial will evaluate a relatively understudied area of menopause - vaginal health and sexual function. This is a 3-arm, randomized, controlled, double-blind, clinical trial among postmenopausal women ages 45-70.

Our primary aim is to evaluate the effectiveness of ultra-low dose vaginal estradiol (Vagifem 10 mcg), non-hormonal hydrophilic non-prescriptive vaginal gel (Replens) and placebo in reducing the Most Bothersome Symptom (MBS) severity. Choices for MBS include vulvovaginal itching, pain, dryness, irritation, or pain with penetration.

Secondary aims include an evaluation of a composite score of vaginal symptoms, sexual function, treatment satisfaction, menopause quality of life, and objective measures of genitourinary atrophy. We will also create a biorepository of vaginal and blood specimens. In a subset of women, we will examine whether treatment response is related to: a) the post-menopausal vaginal microbiome; b) vaginal mucosal inflammation; and c) reproductive hormone profiles. The in-depth focus on the mechanisms associated with postmenopausal vaginal symptoms will use state of the art microbiologic techniques on longitudinally collected biologic specimens and will guide future translational studies.

ELIGIBILITY:
Inclusion Criteria

* Females aged 45-70 years
* 2 or more years since last natural menstrual period, or surgical menopause (bilateral oophorectomy)
* At least 1 vaginal symptom (inside or outside the vagina) reported from the following list, experienced in the past 30 days which is moderate or severe:

  * Dryness at least once a week
  * Itching at least once a week
  * Irritation at least once a week
  * Soreness/Pain at least once a week
  * Pain associated with sexual activity at least once
* Signed informed consent

Exclusion Criteria

* Current unexplained abnormal genital bleeding (or any unevaluated bleeding since menopause)
* Currently pregnant, attempting pregnancy or breast feeding
* Current acute vaginal infection (as indicated by wet mount at V1)
* Pelvic or vaginal surgery in prior 60 days
* Antibiotic use in the past 30 days
* Women under age 55 with endometrial ablation
* Women under age 55 with hysterectomy and at least one ovary
* Current cancer treatment (exception basal or squamous skin cell cancers)
* Current or past thromboembolic disease (pulmonary embolus or deep vein thrombosis, not including thrombophlebitis), myocardial infarction or stroke
* Current severe liver disease
* Current or past breast or endometrial cancer or pre-cancer
* Blood clotting disorder (e.g., Factor V Leiden, prothrombin mutation, protein C, protein or antithrombin deficiency)
* Porphyria
* Current or past lichen sclerosus or lichen planus
* History of adverse reaction to vaginal estrogen or Replens
* Use of any systemic reproductive hormones (hormonal contraception, postmenopausal hormone therapies, SERMS) in the past 2 months
* Use of hormonal contraception in the past year
* Use of any type of vaginal estrogen product (however interested women will be allowed to join the study if they abstain from use during the month preceding enrollment)
* Use of any type of vaginal moisturizer, douche, vaginal prebiotic or probiotic, or soap in the vagina in the past month (however interested women will be allowed to join the study if they abstain from use during the month preceding enrollment)
* Unwilling to abstain from use of any non-study vaginal moisturizer, vaginal estrogen, douche, or soap in the vagina throughout the trial
* Unable to follow instructions, complete questionnaires, or physically unable to place product in the vagina
* Current participation in another drug trial or intervention study
* Chronic vulvo-vaginal symptoms in the 5 years before menopause (defined as a vaginal or vulvar condition requiring more than 4 visits to a health care provider in a given year)

Ages: 45 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine A Guthrie, PhD, Principal Investigator — Fred Hutchinson Cancer Center; Susan D Reed, MD, Principal Investigator — University of Washington; Andrea Z LaCroix, PhD, Principal Investigator — University of California, San Diego; Caroline Mitchell, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - University of Minnesota, Minneapolis, Minnesota
  - Kaiser Permanente Washington Health Research Institute, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
The MsFLASH Data Coordinating Center will perform the statistical analyses for the primary and secondary study results papers. Within a 12-month period after publication of the main study results, the Data Coordinating Center will prepare datasets for public release that include all data elements in the main publication with certain deletions and recoding to protect study subject confidentiality. The public release datasets will include substantial documentation in electronic form, thus allowing external investigators to independently analyze the data.
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Derived] Mitchell CM, Larson JC, Reed SD, Guthrie KA. The complexity of genitourinary syndrome of menopause: number, severity, and frequency of vulvovaginal discomfort symptoms in women enrolled in a randomized trial evaluating treatment for genitourinary syndrome of menopause. Menopause. 2023 Aug 1;30(8):791-797. doi: 10.1097/GME.0000000000002212. Epub 2023 Jul 4. PMID 37402281
- [Derived] Mitchell CM, Larson JC, Crandall CJ, Bhasin S, LaCroix AZ, Ensrud KE, Guthrie KA, Reed SD. Association of Vaginal Estradiol Tablet With Serum Estrogen Levels in Women Who Are Postmenopausal: Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2022 Nov 1;5(11):e2241743. doi: 10.1001/jamanetworkopen.2022.41743. PMID 36374501
- [Derived] Srinivasan S, Hua X, Wu MC, Proll S, Valint DJ, Reed SD, Guthrie KA, LaCroix AZ, Larson JC, Pepin R, Bhasin S, Raftery D, Fredricks DN, Mitchell CM. Impact of Topical Interventions on the Vaginal Microbiota and Metabolome in Postmenopausal Women: A Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2022 Mar 1;5(3):e225032. doi: 10.1001/jamanetworkopen.2022.5032. PMID 35353163
- [Derived] Mitchell CM, Ma N, Mitchell AJ, Wu MC, Valint DJ, Proll S, Reed SD, Guthrie KA, Lacroix AZ, Larson JC, Pepin R, Raftery D, Fredricks DN, Srinivasan S. Association between postmenopausal vulvovaginal discomfort, vaginal microbiota, and mucosal inflammation. Am J Obstet Gynecol. 2021 Aug;225(2):159.e1-159.e15. doi: 10.1016/j.ajog.2021.02.034. Epub 2021 Mar 4. PMID 33675793
- [Derived] Hudson PL, Ling W, Wu MC, Hayward MR, Mitchell AJ, Larson J, Guthrie KA, Reed SD, Kwon DS, Mitchell CM. Comparison of the Vaginal Microbiota in Postmenopausal Black and White Women. J Infect Dis. 2021 Dec 1;224(11):1945-1949. doi: 10.1093/infdis/jiaa780. PMID 33367735
- [Derived] Mitchell CM, Guthrie KA, Larson J, Diem S, LaCroix AZ, Caan B, Shifren JL, Woods NF, Heiman JR, Lindau ST, Reed SD. Sexual frequency and pain in a randomized clinical trial of vaginal estradiol tablets, moisturizer, and placebo in postmenopausal women. Menopause. 2019 Aug;26(8):816-822. doi: 10.1097/GME.0000000000001341. PMID 30994576
- [Derived] Diem SJ, Guthrie KA, Mitchell CM, Reed SD, Larson JC, Ensrud KE, LaCroix AZ. Effects of vaginal estradiol tablets and moisturizer on menopause-specific quality of life and mood in healthy postmenopausal women with vaginal symptoms: a randomized clinical trial. Menopause. 2018 Oct;25(10):1086-1093. doi: 10.1097/GME.0000000000001131. PMID 29738424
- [Derived] Mitchell CM, Reed SD, Diem S, Larson JC, Newton KM, Ensrud KE, LaCroix AZ, Caan B, Guthrie KA. Efficacy of Vaginal Estradiol or Vaginal Moisturizer vs Placebo for Treating Postmenopausal Vulvovaginal Symptoms: A Randomized Clinical Trial. JAMA Intern Med. 2018 May 1;178(5):681-690. doi: 10.1001/jamainternmed.2018.0116. PMID 29554173
- See also: Fred Hutchinson Cancer Research Center website — http://www.fredhutch.org/en/labs/phs/projects/msflash.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Vagifem: One hundred participants will be randomized into the Vagifem® 'active' arm. These women will receive a bottle of Vagifem® tablets (estradiol 10 mcg). One tablet is to be inserted vaginally daily for 2 weeks, then 2 days/week for the remaining 10 weeks of the study.
  Vagifem® tablets contain 10.3 mcg of estradiol hemihydrate equivalent to 10 mcg of estradiol. The excipient (inactive) ingredients are hypromellose, lactose monohydrate, maize starch, and magnesium stearate. Vagifem® comes as a small white film-coated tablet. The coating is made of hypromellose and polyethylene glycol.
  A placebo vaginal gel visually identical composed of inert hydroxyethylcellulose gel (pH adjusted) applied every 3 days over entire 12 weeks.
  Vagifem: One tablet is to be inserted vaginally daily for 2 weeks, then 2 days/week for the remaining 10 weeks of the study.
- Replens: One hundred participants will be randomized into the Replens® 'active' arm. These women will receive a tube containing Replens® vaginal gel. 2.5 gm to be applied vaginally every 3 days over 12 weeks.
  Replens® is a bioadhesive polycarbophil-based moisturizing vaginal gel containing; purified water (vehicle humectant), glycerin (moisturizer), mineral oil (as a moisturizer), polycarbophil and carbomer homopolymer type B (allow the product to stick to the vaginal wall), hydrogenated palm oil glyceride (moisturizer), sorbic acid (preservative, antimicrobial), methylparaben, sodium hydroxide (adjusts pH of product so it is suitable for vaginal use).
  A placebo vaginal tablet visually identical to Vagifem® is inserted daily for 2 weeks, then 2 days/week for remaining 10 weeks.
  Replens: 2.5 gm to be applied vaginally every 3 days over 12 weeks.
  Placebo: Dispensed in visually identical bottle and tablet form.
- Placebo: One hundred participants will be randomized into the 'placebo arm' of the study. This arm is comprised of two placebo preparations; placebo vaginal tablet and placebo vaginal gel applied on the same schedule as 'active' arms.
  The placebo tablet coating and excipient ingredients will be the same as are used for Vagifem®; the coating is made of hypromellose and polyethylene glycol and the excipient (inactive) ingredients are hypromellose, lactose monohydrate, maize starch, and magnesium stearate.
  Placebo vaginal gel. The product is a inert hydroxyethylcellulose gel (pH adjusted).
  Placebo: Dispensed in visually identical bottle and tablet form.
  Placebo: Dispensed in visually identical tube and gel form.
Period: Overall Study
Arm/Group | Vagifem | Replens | Placebo
Started | 102 | 100 | 100
Completed | 100 | 99 | 97
Not Completed | 2 | 1 | 3
Not completed — Withdrawal by Subject | 1 | 0 | 1
Not completed — Lost to Follow-up | 1 | 1 | 1
Not completed — Stopped Follow-up | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vagifem | Replens | Placebo | Total
Number analyzed (Participants) | 102 | 100 | 100 | 302
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (4) | 61 (4) | 61 (4) | 61 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 102 | 100 | 100 | 302
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 87 | 90 | 90 | 267
  Race: African American | 7 | 3 | 2 | 12
  Race: Other / unknown | 8 | 7 | 8 | 23
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Population: 6 participants have missing data on BMI
  kg/m^2
    number analyzed (Participants) | 98 | 100 | 98 | 296
    (all) | 27 (5) | 26 (4) | 26 (6) | 26 (5)
Education [Count of Participants; unit: Participants]
  High school diploma / GED or less | 2 | 3 | 6 | 11
  School after high school | 31 | 27 | 31 | 89
  College graduate | 67 | 70 | 63 | 200
  Missing | 2 | 0 | 0 | 2
Marital status [Count of Participants; unit: Participants]
  Never married | 8 | 2 | 4 | 14
  Divorced or widowed | 10 | 8 | 12 | 30
  Married or like relationship | 83 | 90 | 84 | 257
  Missing | 1 | 0 | 0 | 1
Smoking [Count of Participants; unit: Participants]
  Never | 66 | 67 | 66 | 199
  Past | 31 | 33 | 32 | 96
  Current | 4 | 0 | 2 | 6
  Missing | 1 | 0 | 0 | 1
Alcohol Use [Count of Participants; unit: Participants]
  0 drinks / week | 30 | 31 | 28 | 89
  1-6 drinks / week | 50 | 46 | 53 | 149
  ≥ 7 drinks / week | 21 | 23 | 19 | 63
  Missing | 1 | 0 | 0 | 1
Menopause Quality of Life Questionnaire total [Mean (Standard Deviation); unit: units on a scale] — The Menopause Quality of Life Questionnaire (MENQOL) is a series of 29 questions to assess quality of life in four domains: physical (16 questions), psychosocial (7), sexual (3), and vasomotor (3). Each domain includes occurrence and severity of symptoms; the item scores are averaged for a domain score ranging from 0 (no symptom) to 8 (maximum severity). The four domain scores are then averaged to calculate the total MENQOL score, ranging from 0 (high quality of life) to 8 (low quality of life). Population: 11 participants have missing data for MENQOL total
  units on a scale
    number analyzed (Participants) | 99 | 97 | 95 | 291
    (all) | 3.3 (1.2) | 3.2 (1.1) | 3.3 (1.0) | 3.3 (1.1)
Patient Health Questionnaire 8 depression [Count of Participants; unit: Participants] — The Patient Health Questionnaire (PHQ-8) assesses severity of depression. There are 8 questions, each scored from 0 to 3, that are summed to create a total score ranging from 0 to 24. The scores are categorized as follows: minimal depression (0 to 4), mild depression (5 to 9), moderate depression (10 to 14), moderately severe depression (15 to 19), severe depression (20 to 24).
  Participants
    None (0-4) | 69 | 75 | 69 | 213
    Mild (5-9) | 25 | 22 | 23 | 70
    Moderate - severe (≥10) | 7 | 3 | 8 | 18
    Missing | 1 | 0 | 0 | 1
Generalized Anxiety Disorder Questionnaire 7 [Count of Participants; unit: Participants] — Generalized Anxiety Disorder 7 (GAD-7) assesses generalized anxiety symptoms. It contains 7 questions, each scored from 0 to 3, that are summed to create a total score ranging from 0 to 21. The scores are categorized as follows: minimal GAD (0 to 4), mild GAD (5 to 9), moderate GAD (10 to 14), severe GAD (15 to 21).
  Participants
    None (0-4) | 64 | 75 | 64 | 203
    Mild (5-9) | 25 | 21 | 24 | 70
    Moderate - severe (≥10) | 12 | 4 | 12 | 28
    Missing | 1 | 0 | 0 | 1
Sexually active [Count of Participants; unit: Participants]
  Yes | 81 | 80 | 84 | 245
  No | 20 | 20 | 16 | 56
  Missing | 1 | 0 | 0 | 1
Female Sexual Distress Scale-Revised, item 1, distressed about sex life [Count of Participants; unit: Participants]
  Never / rarely | 15 | 12 | 18 | 45
  Occasionally | 33 | 33 | 33 | 99
  Frequently / always | 53 | 54 | 49 | 156
  Missing | 1 | 1 | 0 | 2
Female Sexual Function Index total [Mean (Standard Deviation); unit: units on a scale] — The Female Sexual Function Index (FSFI) assesses sexual functioning in women. It consists of 19 questions grouped into 6 domains: desire (2 questions), arousal (4), lubrication (4), orgasm (3), satisfaction (3), and pain (3). Each domain score ranges from a low value between 0 and 1.2 (varies by domain) and a high value of 6. The domain scores are summed to calculate the total FSFI score (range 2-36), with high scores indicating better sexual function. Population: 50 participants have missing data on FSFI total
  units on a scale
    number analyzed (Participants) | 81 | 86 | 85 | 252
    (all) | 15.2 (539) | 15.2 (6.5) | 16.1 (6.6) | 15.5 (6.4)
Vaginal pH [Count of Participants; unit: Participants]
  ≤ 5 | 18 | 12 | 9 | 39
  > 5 | 81 | 87 | 90 | 258
  Missing | 3 | 1 | 1 | 5
Vaginal maturation index [Count of Participants; unit: Participants]
  ≤ 5% superficial cells | 86 | 78 | 81 | 245
  > 5% superficial cells | 6 | 11 | 7 | 24
  Missing | 10 | 11 | 12 | 33
Most bothersome symptom [Count of Participants; unit: Participants]
  Vulvar and/or vaginal itching | 10 | 4 | 6 | 20
  Vulvar and/or vaginal pain | 5 | 7 | 2 | 14
  Vaginal dryness | 23 | 17 | 23 | 63
  Vulvar and/or vaginal irritation | 7 | 4 | 8 | 19
  Pain with vaginal penetration | 54 | 68 | 60 | 182
  Missing | 3 | 0 | 1 | 4
Self-reported health [Count of Participants; unit: Participants]
  Excellent | 26 | 27 | 20 | 73
  Very good | 41 | 55 | 47 | 143
  Good | 33 | 15 | 30 | 78
  Fair / poor | 1 | 3 | 3 | 7
  Missing | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Most Bothersome Symptom (MBS) Severity
Description: Mean change from baseline to 12 weeks in the severity of the MBS on a scale of 0-3, better to worse.
Time Frame: Baseline, Week 4, Week 12
Population: Analysis includes participants with MBS data at baseline and either week 4 or 12.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Vagifem | Replens | Placebo
Number analyzed (Participants) | 97 | 99 | 98
units on a scale
  Week 4 minus baseline | -1.2 [-1.4 to -1.0] | -1.0 [-1.2 to -0.8] | -0.2 [-0.5 to 0.1]
  Week 12 minus baseline | -1.4 [-1.6 to -1.2] | -1.2 [-1.4 to -1.0] | -1.3 [-1.5 to -1.1]
Statistical Analysis 1: Comparison: Vagifem vs Placebo; Test type: Superiority; p = 0.25, Regression, Linear — P-values from active treatment vs. placebo contrasts in a repeated measures linear model of outcome as a function of treatment arm, clinical site, week, and baseline outcome. The a priori threshold for statistical significance was 0.025; Robust standard errors were calculated using generalized estimating equations to account for within-participant correlation between repeated measures
Statistical Analysis 2: Comparison: Replens vs Placebo; Test type: Superiority; p = 0.31, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]

2. Secondary Outcome: Vaginal Symptoms Index
Description: Mean change from baseline to 12 weeks in composite Vaginal Symptoms Index (VSI).
  The VSI is a Modified Bachman scale measuring vulvovaginal itching, dryness, irritation, soreness, and pain with sexual activity among sexually active women, each rated 0=none to 3=severe, and then averaged for a total score of 0-3.
Time Frame: Baseline, Week 4, Week 12
Population: Analysis includes participants with VSI data at baseline and either week 4 or 12.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Vagifem | Replens | Placebo
Number analyzed (Participants) | 100 | 99 | 99
units on a scale
  Week 4 minus baseline | -0.7 [-0.8 to -0.5] | -0.5 [-0.7 to -0.4] | -0.6 [-0.8 to -0.5]
  Week 12 minus baseline | -0.9 [-1.1 to -0.8] | -0.7 [-0.9 to -0.6] | -0.9 [-1.0 to -0.7]
Statistical Analysis 1: Comparison: Vagifem vs Placebo; Test type: Superiority; p = 0.99, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Replens vs Placebo; Test type: Superiority; p = 0.05, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]

3. Secondary Outcome: Female Sexual Function Index
Description: Female Sexual Function Index (FSFI); Evaluate dyspareunia, sexual function and distress. A composite score from 2 (not sexually active and no desire) to 36 and 6 domains.
Time Frame: Baseline, Week 4, Week 12
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Vagifem | Replens | Placebo
Number analyzed (Participants) | 70 | 81 | 82
units on a scale
  Week 4 minus baseline | 3.1 [1.5 to 4.7] | 2.9 [1.7 to 4.1] | 3.2 [1.8 to 4.7]
  Week 12 minus baseline | 5.4 [4.0 to 6.9] | 3.1 [1.7 to 4.5] | 4.5 [2.8 to 6.1]
Statistical Analysis 1: Comparison: Vagifem vs Placebo; Test type: Superiority; p = 0.64, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Replens vs Placebo; Test type: Superiority; p = 0.17, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]

4. Secondary Outcome: Treatment Satisfaction
Description: Likert Scale 0 = no to 10 = complete satisfaction.
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vagifem | Replens | Placebo
Number analyzed (Participants) | 98 | 99 | 95
units on a scale | 8.6 (2.6) | 7.7 (3.2) | 8.1 (3.0)

5. Secondary Outcome: Patient Benefit Evaluation
Description: Patient Benefit Evaluation: Overall, do you believe that you experienced a meaningful benefit from the study medication? (Yes/No).
Time Frame: Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | Vagifem | Replens | Placebo
Number analyzed (Participants) | 102 | 100 | 100
Participants
  Yes | 79 | 58 | 62
  No | 20 | 41 | 34
  Missing | 3 | 1 | 4
Statistical Analysis 1: Comparison: Vagifem vs Placebo; Test type: Superiority; p = 0.02, Chi-squared — p-value calculation includes 195 participants with known responses at week 12

6. Secondary Outcome: pH
Description: Objective measures of genitourinary atrophy: pH (<5 or >5) at week 12
Time Frame: Week 12
Population: Sample includes 247 participants with pH > 5 at baseline and non-missing data on pH at week 12
Measure: Count of Participants; unit: Participants
Arm/Group | Vagifem | Replens | Placebo
Number analyzed (Participants) | 78 | 85 | 84
Participants
  Week 12 pH > 5 | 42 | 77 | 74
  Week 12 pH ≤ 5 | 36 | 8 | 10
Statistical Analysis 1: Comparison: Vagifem vs Placebo; Test type: Superiority; p < 0.001, Chi-squared
Statistical Analysis 2: Comparison: Replens vs Placebo; Test type: Superiority; p = 0.60, Chi-squared

7. Secondary Outcome: Vaginal Maturation Index
Description: Objective Measures of Genitourinary Atrophy: Vaginal Maturation Index (VMI) described by % parabasal, intermediate, and superficial cells (≤ 5% or >5% superficial cells) at week 12
Time Frame: Week 12
Population: Sample includes 223 participants with VMI ≤ 5% superficial cells at baseline and non-missing VMI data at week 12
Measure: Count of Participants; unit: Participants
Arm/Group | Vagifem | Replens | Placebo
Number analyzed (Participants) | 79 | 73 | 71
Participants
  Week 12 VMI ≤ 5% | 34 | 65 | 63
  Week 12 VMI > 5% | 45 | 8 | 8
Statistical Analysis 1: Comparison: Vagifem vs Placebo; Test type: Superiority; p < 0.001, Chi-squared
Statistical Analysis 2: Comparison: Replens vs Placebo; Test type: Superiority; p = 0.95, Chi-squared

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for each participant from randomization through the 12-week visit.
Arm/Group | Vagifem | Replens | Placebo
All-Cause Mortality (participants affected / at risk) | 0/102 | 0/100 | 0/100
Serious Adverse Events (participants affected / at risk) | 3/102 | 1/100 | 1/100
Other Adverse Events (participants affected / at risk) | 26/99 | 22/99 | 24/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vagifem (N=102) | Replens (N=100) | Placebo (N=100)
Hospitalization for dehydration (Gastrointestinal disorders) | 0 | 1 | 0 — Admitted to hospital for ongoing gastrointestinal symptoms. Admitted again 6 days later with dehydration diagnosis.
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 — Lobular carcinoma in left breast
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 — Lymphoma confirmed by lab tests
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 — Infiltrating ductal carcinoma left breast
Hospitalization for back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 — Participant reported increasing back pain, worsening spinal stenosis, required surgery
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Vagifem (N=99) | Replens (N=99) | Placebo (N=99)
Increased vaginal secretions (Reproductive system and breast disorders) | 14/92 | 16 | 14/96 — Counted in participants who did not report moderate-severe vaginal secretions at baseline
Vaginal itching (Reproductive system and breast disorders) | 6/75 | 6/79 | 6/84 — Counted in participants who did not report moderate-severe vaginal itching at baseline
Breast tenderness (Reproductive system and breast disorders) | 3/97 | 0/98 | 2/96 — Counted in participants who did not report moderate-severe breast tenderness at baseline
Vaginal spotting or bleeding (Reproductive system and breast disorders) | 0 | 1 | 0 — Counted in participants who did not report moderate-severe vaginal spotting or bleeding at baseline
Skin rash outside the vagina (Skin and subcutaneous tissue disorders) | 4/96 | 0/97 | 1/97 — Counted in participants who did not report moderate-severe skin rash outside the vagina at baseline
Body rash (Skin and subcutaneous tissue disorders) | 2/95 | 1/97 | 5/98 — Counted in participants who did not report moderate-severe body rash at baseline

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-11-01): https://cdn.clinicaltrials.gov/large-docs/02/NCT02516202/Prot_SAP_000.pdf
  • Informed Consent Form (2016-11-01): https://cdn.clinicaltrials.gov/large-docs/02/NCT02516202/ICF_001.pdf